CLINICAL TRIAL: NCT00649961
Title: Melatonin As A Novel Neuroprotectant In Preterm Infants- Dosage Study
Acronym: MIND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: British Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR0970 (MIND); 2007-007156-33 (EudraCT Number)
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Premature Birth; Brain Injury
Keywords: Premature Birth; Brain injury; Neuroprotection; Melatonin; Pharmacokinetics
MeSH Terms: conditions — Premature Birth; Brain Injuries | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Melatonin Open Label Single Arm (Experimental): Infants born less than 31 weeks gestation who are less than 7 days old
  Interventions: Drug: Melatonin injection

INTERVENTIONS:
Drug: Melatonin injection — A single intravenous infusion of melatonin will be given to each infant over 6 hours so that successive groups will receive increasing doses until the correct dose for age is found.
  Based on the pharmacokinetics and clearance of melatonin in adults an approximate dose has been calculated. The starting dose of melatonin will be 0.1 microgram/kg/hr to be given over 6 hours intravenously. The range of expected dose is 0.1-0.5 microgram/kg/hr.
  Other Names: CAS-73314

SUMMARY:
Preterm babies are at risk of brain injury. Melatonin, a naturally occurring hormone, may reduce this risk. The unborn baby receives melatonin from the mother but following premature delivery there maybe a period of prolonged melatonin deficiency. This deficiency may be harmful because studies suggest that melatonin is important in protecting the brain and reducing the risk of brain injury after preterm birth. The purpose of this study is to find the ideal dose of melatonin to give to preterm babies. We intend to study a total of 24 babies less than 31 weeks gestation and who are less than 7 days old.

DETAILED DESCRIPTION:
PURPOSE OF THE STUDY AND OBJECTIVES The overall purpose is to investigate whether melatonin, on achieving adult maternal peak blood levels in preterm infants, will reduce brain injury and white matter disease as defined by specialised magnetic resonance imaging (MRI) at term. Before testing this hypothesis in a clinical trial, the dose of melatonin required to achieve the desired concentration in preterm infants needs to be determined. This data will be used in the clinical double blinded randomised trial for which a separate application will be made to the ethics committee.

The principal research objective in this study is to determine the dose required to achieve physiological melatonin blood levels in the preterm infants similar to that of the mother. Secondary objective is to define the pharmacokinetic profile of melatonin in preterm infants.

STUDY DESIGN AND METHODOLOGY The proposed clinical trial is a single dose, open label, dose escalation pharmacokinetic study in preterm infants less than 31weeks gestation to achieve adult peak blood concentrations of melatonin (200-250 pmol/L).

The trial will be a multi centre study based in the Neonatal Intensive Care Units in UK.

TREATMENT A single intravenous infusion of melatonin will be given to each infant over 6 hours once in the first 7 days of life. The starting dose is 0.1 microgram/kg/hr which will be increased or decreased incrementally in subsequent groups of infants until the desired melatonin concentration is achieved.

DURATION The duration of treatment will be 6 hours only.

INVESTIGATIONS Pharmacokinetic assessment will be performed on the blood and urine samples will be collected 2 hourly at various timepoints.

STATISTICAL ANALYSIS Pharmacokinetic assessment will be done using appropriate software.

ELIGIBILITY:
Inclusion Criteria:

* Infants born less than 31 weeks gestation who are less than 7 days old, after parental consent for participation will be included in the study.

Exclusion Criteria:

* Those with major congenital malformation, or cystic periventricular leucomalacia (cPVL) or haemorrhagic parenchymal infarcts (HPI) on cranial ultrasonography prior to enrolment will be excluded from the study.

Ages: 23 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Edwards, FRCPCH, Principal Investigator — Imperial College London; Denis Azzopardi, FRCPCH, Principal Investigator — Imperial College London; Nazakat Merchant, MRCPCH, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Royal Bolton Hospital, Bolton
  - Imperial College Healthcare NHS Trust, London

REFERENCES:
- [Background] Jan JE, Wasdell MB, Freeman RD, Bax M. Evidence supporting the use of melatonin in short gestation infants. J Pineal Res. 2007 Jan;42(1):22-7. doi: 10.1111/j.1600-079X.2006.00398.x. PMID 17198535
- [Background] Volpe JJ. Cerebral white matter injury of the premature infant-more common than you think. Pediatrics. 2003 Jul;112(1 Pt 1):176-80. doi: 10.1542/peds.112.1.176. No abstract available. PMID 12837883
- [Background] Wood NS, Marlow N, Costeloe K, Gibson AT, Wilkinson AR. Neurologic and developmental disability after extremely preterm birth. EPICure Study Group. N Engl J Med. 2000 Aug 10;343(6):378-84. doi: 10.1056/NEJM200008103430601. PMID 10933736
- See also: Medicines for Children Regulatory Network- adopted study — http://www.mcrn.org.uk
- See also: UK Medical Research Council- funder for the study — http://www.mrc.ac.uk

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We conducted an open label dose ranging study between May 2010 and December 2010 in 3 neonatal intensive care units in the UK.
Pre-assignment Details: Infants born less than 31 weeks gestation and less than 7 days old were eligible for the study, although those with: major congenital malformation; or cystic periventricular leucomalacia or haemorrhagic parenchymal infarcts on cranial enrolment were excluded.
Groups:
- Melatonin Open Label Single Arm: Open label single arm study, infant born less than 31 weeks gestation and less than 7 days old
Period: Overall Study
Arm/Group | Melatonin Open Label Single Arm
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Infants born at less than 31 weeks gestation and less than 7 days after birth
Groups:
- Single Arm: Open label dose finding study in infants born before 31 weeks gestation and less than 7 days of age
Arm/Group | Single Arm
Number analyzed (Participants) | 18
Age, Customized [Median (Full Range); unit: weeks]
  Gestation at birth | 26.63 [24.71 to 30.28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Region of Enrollment [Number; unit: participants]
  United Kingdom | 18

OUTCOME MEASURES:

1. Primary Outcome: To Find the Dose of Melatonin Required to Achieve Physiological Blood Levels in the Preterm Infants Similar to That of the Mother.
Time Frame: 6 months
Measure: Median (Full Range); unit: pg/ml
Groups:
- Single Arm: open label dose finding study
Arm/Group | Single Arm
Number analyzed (Participants) | 18
pg/ml | 203.3 [160 to 220]

ADVERSE EVENTS:
Time Frame: 6 month
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less